CLINICAL TRIAL: NCT03374241
Title: A First-in-human Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics After Single Ascending Dose of HM15211(Efocipegtrutide) in Healthy Obese Subjects
Brief Title: A First-in-human Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of HM15211(Efocipegtrutide)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: HM-TRIA-101
Record Dates: First submitted 2017-12-12; First posted 2017-12-15 (Actual); Results first posted 2024-05-17 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Experimental): HM15211 or Placebo (single dose, subcutaneous injection)
  Interventions: Biological: HM15211 or Placebo
- Cohort 2 (Experimental): HM15211 or Placebo (single dose, subcutaneous injection)
  Interventions: Biological: HM15211 or Placebo
- Cohort 3 (Experimental): HM15211 or Placebo (single dose, subcutaneous injection)
  Interventions: Biological: HM15211 or Placebo
- Cohort 4 (Experimental): HM15211 or Placebo (single dose, subcutaneous injection)
  Interventions: Biological: HM15211 or Placebo
- Cohort 5 (Experimental): HM15211 or Placebo (single dose, subcutaneous injection)
  Interventions: Biological: HM15211 or Placebo

INTERVENTIONS:
Biological: HM15211 or Placebo — Long-acting tri-agonist

SUMMARY:
Single ascending dose of HM15211 in healthy obese subjects.

DETAILED DESCRIPTION:
A First-in-human study to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics after single ascending dose of HM15211 in healthy obese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects must be non-pregnant and non-lactating

Exclusion Criteria:

* Participation in an investigational study within 30 days prior to dosing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2018-09-14 (Actual); Study Completion 2018-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hanmi Pharmaceuticals, Study Director — Hanmi Pharmaceuticals
Locations (1):
- Hanmi Investigative Site, Chula Vista, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: HM15211 0.01 mg/kg
- Cohort 2: HM15211 0.02 mg/kg
- Cohort 3: HM15211 0.04 mg/kg
- Cohort 4: HM15211 0.08 mg/kg
- Cohort 5: HM15211 0.12 mg/kg
- Placebo: Placebo matched to the volume of the dose of HM15211
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Placebo
Started | 6 | 6 | 6 | 7 | 6 | 10
Completed | 6 | 6 | 5 | 5 | 5 | 10
Not Completed | 0 | 0 | 1 | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Population: all randomized subjects (total 41)
Groups:
- Cohort 1 Active: HM15211 0.01 mg/kg
- Cohort 2 Active: HM15211 0.02 mg/kg
- Cohort 3 Active: HM15211 0.04 mg/kg
- Cohort 4 Active: HM15211 0.08 mg/kg
- Cohort 5 Active: HM15211 0.12 mg/kg
- Total: Total of all reporting groups
Arm/Group | Cohort 1 Active | Cohort 2 Active | Cohort 3 Active | Cohort 4 Active | Cohort 5 Active | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 6 | 10 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 6 | 7 | 6 | 10 | 41
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.0 (14.34) | 36.3 (11.78) | 54.0 (6.13) | 49.7 (11.06) | 43.8 (13.53) | 47.4 (6.55) | 45.7 (11.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 2 | 4 | 2 | 5 | 20
  Male | 3 | 2 | 4 | 3 | 4 | 5 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 5 | 1 | 3 | 4 | 4 | 18
  Not Hispanic or Latino | 5 | 1 | 5 | 4 | 2 | 6 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Black or African American | 2 | 1 | 4 | 1 | 0 | 4 | 12
  White | 4 | 5 | 2 | 5 | 6 | 5 | 27
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 7 | 6 | 10 | 41

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: An adverse event is any undesirable and unintended medical event occurring to a subject in a clinical study, whether or not related to the investigational products
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Active | Cohort 2 Active | Cohort 3 Active | Cohort 4 Active | Cohort 5 Active | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 6 | 10
Participants | 3 | 2 | 3 | 7 | 4 | 7

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Cohort 1 Active | Cohort 2 Active | Cohort 3 Active | Cohort 4 Active | Cohort 5 Active | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/7 | 0/6 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/7 | 0/6 | 0/10
Other Adverse Events (participants affected / at risk) | 3/6 | 2/6 | 3/6 | 7/7 | 4/6 | 7/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 Active (N=6) | Cohort 2 Active (N=6) | Cohort 3 Active (N=6) | Cohort 4 Active (N=7) | Cohort 5 Active (N=6) | Placebo (N=10)
GI disorders (Gastrointestinal disorders) | 0 | 0 | 1 | 4 | 4 | 1
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Eye disorders (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Infections and infestations (Infections and infestations) | 1 | 0 | 0 | 0 | 2 | 0
Injury, poisoning and procedural (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal and connective tissue (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0 | 1 | 0
Nervous system disorders (Nervous system disorders) | 0 | 1 | 0 | 4 | 2 | 2
Renal and urinary disorders (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Respiratory, thoracic and mediastinal (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
General disorders and administration (General disorders) | 2 | 1 | 1 | 2 | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-04-06): https://cdn.clinicaltrials.gov/large-docs/41/NCT03374241/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-17): https://cdn.clinicaltrials.gov/large-docs/41/NCT03374241/SAP_001.pdf